CLINICAL TRIAL: NCT03012893
Title: Identification of the C7 Vertebral Level; Evaluations of Two Sonographic Methods Using a Transverse Scan of the C7 Transverse Process and a Sagittal Scan of the First Rib.
Brief Title: Identification of C7; Evaluations of 2 Sonographic Methods Using a Transverse and a Sagittal Scan.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 554/2559(EC2)
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Breastcancer
Keywords: ultrasonography to identify C7 spinous process

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ultrasound transverse scan (Experimental): Transvers scan by identifying the C7 transvers process using vertebral artery and absence of anterior tubercle as a landmark and then scan back following articular process, lamina and then find out the spinous process of C7
  Interventions: Device: Ultrasound transverse scan
- Ultrasound sagittal scan (Experimental): Sagittal scan by identifying the first and second ribs and scan medially to depict the C7 transvers process.
  Interventions: Device: Ultrasound sagittal scan
- Floroscopic technique (Active Comparator): Fluoroscopy image will do on lateral view including all cervical spines and upper thoracic spines. C7 spinous process will be identified by counting down from C1 vertebral body and spinous process.
  Interventions: Procedure: Fluoroscopic technique

INTERVENTIONS:
Device: Ultrasound sagittal scan — Convex transducer will be placed at patient's neck using paramedian sagittal scan and pointing toward the chest apex aiming to identify the first rib. Then move the transducer medially to identify the transverse process along with identify C7 transverse process will appear on the image as a hyperechoic shadow without continue to the rib laterally. Place the C7 spinous process on the midpoint of the probe and the spinous process correspondence to the midline will be marked as C7.
  Arms: Ultrasound sagittal scan
Device: Ultrasound transverse scan — Linear transducer will be placed at patient's lateral neck using transverse scan. The unique characteristic of sonography of transvers process of C6 and C7 will be used to identify the transverse process of C6 and C7. C6 transverse process has a very prominence anterior tubercle (known as Chassaignac tubercle). While anterior tubercle of C7 is absent. After identifying the C7 transverse process, simultaneously the color Doppler mode will be activated to identify the vertebral artery for double confirmation.
  Arms: Ultrasound transverse scan
Procedure: Fluoroscopic technique — C7 spinous process will be identified by counting down from C1 vertebral body and spinous process.
  Arms: Floroscopic technique

SUMMARY:
To determine the accuracy of two techniques (transverse scan and sagittal scan) using ultrasonography to identify C7 spinous process compare to the fluoroscope (standard technique)

DETAILED DESCRIPTION:
To identify the accurate level of upper thoracic spine is essential maneuver during breast surgery and axillary node dissection. Palpation C7 spinous process is most common technique using to identify the level. However, the accuracy was lower than 50%. Ultrasonography has been investigated to identify the cervical nerve roots by differentiating the transvers process of C6 and C7. However, there was no study on the accuracy of using ultrasound to identify cervical spine level before.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer, age >/= 18

Exclusion Criteria:

* previous cervical spine surgery, cervical spine deformity, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
the accuracy of identify C7 spinous process | 1 day
  the accuracy of two techniques (transverse scan and sagittal scan) using ultrasonography to identify C7 spinous process compare to the fluoroscope (standard technique)

IPD SHARING:
Plan to Share IPD: No